CLINICAL TRIAL: NCT01658722
Title: A Phase 3b Study of Subjects With Alzheimer's Disease Who Discontinued Treatment in Bapineuzumab Phase 3 Clinical Studies (ELN115727-301/302/351) or Who Completed Studies ELN15727-301 and 302 But Did Not Enroll in Study ELN115727-351
Brief Title: Retrieval of Patient Information After Discontinuation
Acronym: RAPID
Status: Terminated | Type: Observational
Sponsor: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: AAB-001-ALZ-3300
Record Dates: First submitted 2012-03-12; First posted 2012-08-07 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2012-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — bapineuzumab

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Observational: Long term follow-up
  Interventions: Drug: Bapineuzumab

INTERVENTIONS:
Drug: Bapineuzumab

SUMMARY:
A Phase 3b, Study of Subjects With Alzheimer's Disease Who Discontinued Treatment in Bapineuzumab Phase 3 Clinical Studies (ELN115727-301/302/351) or Who Completed Studies ELN115727-301 and 302 but did not Enroll in Study ELN115727-351.

ELIGIBILITY:
1. Signed, dated, and written informed consent obtained from the subject and/or the subject's legally acceptable representative (LAR, if applicable) in accordance with local regulations.
2. Signed, dated, and written informed consent, obtained from the subject's caregiver in accordance with local regulations.
3. Subject must have participated in the Study 301, 302, or 351 and have received at least 1 dose of study treatment (bapineuzumab or placebo).
4. Subject must have been off treatment for at least 12 months prior to Visit 1.
5. Subjects must have a primary caregiver for the duration of the study.
6. Subject's caregiver must have the ability to assess the subject and answer questions over the phone.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Alzheimer's disease who discontinued treatment in bapineuzumab Phase 3 clinical studies (ELN115727-301/302/351) or who completed studies ELN115727-301 or 302 but did not enroll in study ELN115727-351
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Dependence Scale | 4 years
  Caregiver's assessment of a patient's need for assistance